CLINICAL TRIAL: NCT07139145
Title: Effect of Adding Progressive Muscle Relaxation to Physical Therapy Program on Fatigue, Mobility and Stress Among Traumatic Lower Limb Amputees in Gaza Strip
Brief Title: Effect of Adding Progressive Muscle Relaxation to Physical Therapy Program on Fatigue, Mobility and Stress Among Individuals With Traumatic Lower Limb Amputation in the Gaza Strip
Acronym: PMR-AMP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marah Radi (Other)
Responsible Party: Sponsor-Investigator, Marah Radi, Master's Student, Faculty of Applied Medical Sciences, Al-Azhar University - Gaza, Al-Azhar University
Organization: Al-Azhar University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PHRC/HC/1251/25
Record Dates: First submitted 2025-08-17; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Traumatic Lower Limb Amputation; Fatigue; Mobility Impairment; Psychological Stress
Keywords: Progressive Muscle Relaxation (PMR); Physiotherapy; Rehabilitation; Fatigue; Mobility; Stress; Weight-Bearing Symmetry; Gaza Strip; Amputees; Randomized Controlled Trial (RCT)
MeSH Terms: conditions — Fatigue; Stress, Psychological | interventions — Autogenic Training

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocated in a 1:1 ratio to either an intervention group (standard physiotherapy plus Progressive Muscle Relaxation) or a control group (standard physiotherapy alone). The trial will follow a parallel-group design, with outcomes assessed at baseline, post-intervention (6 weeks), and follow-up (8 weeks).
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental - Physiotherapy + Progressive Muscle Relaxation (PMR) (Experimental): Participants receive a 6-week standard physiotherapy program combined with Progressive Muscle Relaxation (PMR). Physiotherapy includes warm-up, weight-bearing training, balance training, gait training, and functional activities, delivered twice weekly. PMR sessions last 20 minutes, twice weekly, and involve systematic tensing/relaxing of major muscle groups, diaphragmatic breathing, and visualization techniques adapted for amputees.
  Interventions: Behavioral: Progressive Muscle Relaxation + Standard Physiotherapy
- Active Comparator - Standard Physiotherapy Only (Active Comparator): Participants receive the same 6-week standard physiotherapy program as the intervention group (warm-up, weight-bearing training, balance training, gait training, and functional activities, twice weekly) but without Progressive Muscle Relaxation.
  Interventions: Behavioral: Standard Physiotherapy

INTERVENTIONS:
Behavioral: Progressive Muscle Relaxation + Standard Physiotherapy — Standard physiotherapy exercises plus PMR sessions. PMR is gradually transitioned from therapist-guided to self-directed practice across the 6 weeks.
  Arms: Experimental - Physiotherapy + Progressive Muscle Relaxation (PMR)
Behavioral: Standard Physiotherapy — Participants receive a 6-week standard physiotherapy program delivered twice weekly. Sessions include warm-up, weight-bearing training, balance exercises, gait training, and functional activities. The protocol focuses on improving mobility, weight-bearing capacity, balance, and functional independence. No Progressive Muscle Relaxation or additional behavioral techniques are included.
  Arms: Active Comparator - Standard Physiotherapy Only

SUMMARY:
Lower limb amputation is a life-altering condition with profound physical and psychological consequences, including fatigue, impaired mobility, stress, and asymmetrical weight-bearing. These challenges are particularly severe in conflict-affected settings like the Gaza Strip, where access to rehabilitation services is limited.

This study aims to evaluates the effect of adding Progressive Muscle Relaxation (PMR), a simple and cost-effective relaxation technique, to standard physical therapy on Fatigue, mobility, weightbearing distribution and stress outcomes among adults with unilateral traumatic lower limb amputation in Gaza.

Study design:

RCT with 60 participants will be randomly assigned to either (1) a control group receiving standard physiotherapy or (2) an intervention group receiving standard physiotherapy plus PMR.

Outcomes will be measured using validated instruments: Fatigue Severity Scale (FSS), 2-Minute Walk Test (2MWT), Perceived Stress Scale (PSS-10), and dual bathroom scale method for weight-bearing distribution. Assessments will be conducted at baseline, post-intervention (6 weeks), and follow-up (8 weeks).

The study aims to determine whether integrating PMR into rehabilitation improves fatigue reduction, functional mobility, stress management, and weight-bearing symmetry compared to physiotherapy alone. Findings will contribute to evidence-based rehabilitation strategies for amputees in low-resource, high-stress environments.

DETAILED DESCRIPTION:
This study protocol addresses the multidimensional challenges faced by individuals with traumatic lower limb amputation in the Gaza Strip, a conflict-affected region with limited access to rehabilitation. Amputees often experience persistent fatigue, impaired mobility, asymmetrical weight-bearing, and high psychological distress. Standard physical therapy primarily focuses on physical recovery, while psychosocial rehabilitation is often overlooked.

Rationale:

Progressive Muscle Relaxation (PMR) is a structured mind-body technique that systematically tenses and relaxes muscle groups to reduce stress and physical tension. Evidence from other populations, including patients with cancer, chronic illnesses, and stroke, has shown PMR to be effective in reducing fatigue, anxiety, stress, and improving functional performance. However, its use in amputee rehabilitation-particularly in conflict settings-remains underexplored.

Study Objectives:

General Objective: To evaluate the effect of integrating PMR with physiotherapy program on Fatigue, mobility, weightbearing distribution and stress among individuals with traumatic lower limb amputation.

Study Design:

Randomized controlled trial (RCT) with 60 participants allocated to intervention (PMR + physiotherapy) or control (physiotherapy alone) groups using block randomization and concealed allocation.

Outcome Measures:

Fatigue (FSS), mobility (2MWT), Stress (PSS-10), weight-bearing symmetry (dual scale method).

Assessment Timeline: Baseline (week 0), post-intervention (week 6), and follow-up (week 8).

Sample Size: 60 participants (30 per group), based on power analysis accounting for attrition.

Data Analysis: Descriptive statistics, paired t-tests, independent t-tests, and repeated-measures ANOVA. Intention-to-treat analysis will be applied.

Ethics: Approval is obtained from the Helsinki Committee and the Artificial Limbs and Polio Center (ALPC). Informed consent will be secured, confidentiality maintained, and adverse events monitored.

Expected Impact:

This study will provide the first randomized evidence on the effectiveness of PMR in traumatic amputee rehabilitation within Gaza. It is expected that adding PMR to physiotherapy will significantly reduce fatigue and stress, improve mobility, and enhance weight-bearing symmetry compared to physiotherapy alone. Results will inform rehabilitation protocols in low-resource, conflict-affected settings and may guide future policy and practice for amputee care.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 59 years.
* Unilateral traumatic trans-femoral/transtibial amputation.
* Post prosthetic fitting.

Exclusion Criteria:

* Severe comorbidities (e.g., uncontrolled cardiovascular disease).
* Severe cognitive impairment or mental illness.
* Recent orthopaedic surgery (<3 months)

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2025-11-15 (Estimated); Study Completion 2026-02-26 (Estimated)

PRIMARY OUTCOMES:
Fatigue Level | Baseline, 6 weeks post-intervention and 8 weeks follow up
  Assessed using the Fatigue Scale-2, measuring perceived physical and mental fatigue. Scores quantify fatigue severity.
Mobility | Baseline, 6 weeks post-intervention and 8 weeks Follow up
  Measured using the 2-Minute Walk Test (2MWT) to assess distance walked in meters.
Stress Level | Baseline, 6 weeks post-intervention and 8 weeks following
  Assessed with a validated Perceived Stress Scale measuring psychological stress
Weight-Bearing distribution | Baseline, 6 weeks post-intervention and 8 weeks following
  Measured using a dual bathroom scale during standing tasks to assess weight-bearing capacity.

CONTACTS AND LOCATIONS:
Overall Officials: Mosab Aldabbas, PhD, Study Chair — Al-Azhar University, Gaza Strip
Locations (1):
- Artificial Limb & Polio Center (ALPC), Gaza, Gaza, Palestinian Territories

IPD SHARING:
Plan to Share IPD: No
individual participant data will not be shared. Data will be kept confidential and used solely for the purposes of this study